CLINICAL TRIAL: NCT01340924
Title: Key Determinants of Type 2 Diabetes Prevention Among Women With a History of Gestational Diabetes Mellitus
Brief Title: Relationship Between Gestational Diabetes and Type 2 Diabetes
Acronym: GDM
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Laval University (Other)
Responsible Party: Principal Investigator, Julie Robitaille, Assistant Professor, Laval University
Other Study IDs: GDM
Record Dates: First submitted 2011-03-15; First posted 2011-04-25 (Estimated); Last update posted 2022-04-08 (Actual); Status verified 2022-04

CONDITIONS: Gestational Diabetes; Type 2 Diabetes
Keywords: Gestational diabetes; Type 2 diabetes
MeSH Terms: conditions — Diabetes, Gestational; Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood; serum; white cell.
Oversight: Data Monitoring Committee: No

SUMMARY:
The overall objective of this research project is to study the impact of preventive practices on the T2D-related risk profile among women with and without prior GDM and their children exposed and unexposed to GDM.

DETAILED DESCRIPTION:
Type 2 diabetes (T2D) is a growing public health problem owing to its prevalence as well as its high morbidity and mortality rates. The identification of high-risk populations is of great importance particularly because the onset of T2D can be prevented or delayed by lifestyle modifications. Among high-risk populations, women with previously diagnosed gestational diabetes mellitus (GDM) are at particularly high risk of developing T2D. The success in reducing the occurrence of T2D among women with previous GDM could be achieved only if appropriate preventive measures are undertaken. According to the American Diabetes Association (ADA) and the Canadian Diabetes Association (CDA), lifestyle modifications aimed at reducing body weight and increasing physical activity are recommended and women are encouraged to be breastfeeding their infants. Certain factors have been suggested as determinants of behavioral practices in women with prior GDM including cognitive and environmental factors. A better understanding of these issues is essential for developing effective preventive strategies and possibly reducing the prevalence of T2D in the population. Moreover, in utero exposure to maternal impaired glucose tolerance or diabetes may increase the risk of developing overweight or diabetes in offspring. Since March 2012 we thus test the presence of childhood metabolic alterations predictive of future T2D in GDM-exposed and unexposed offspring and investigate environmental factors during the postnatal period that are associated with prevention of metabolic alterations.

ELIGIBILITY:
Inclusion Criteria:

* Women aged ≥18 years with or without a diagnosis of GDM in the past 3-12 years and their children.

Exclusion Criteria:

* Pregnant women, women with type 1 diabetes.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In order to avoid selection biases, we plan to recruit 450 women with a history of GDM through administrative data from the Régie de l'assurance maladie du Québec (RAMQ) and children of those mothers.
  We plan to recruit 125 women without history of GDM through mail sent to students and employees of local university and children of those mothers.
Sampling Method: Non-Probability Sample
Enrollment: 450 (Estimated)
Dates: Start 2009-09; Primary Completion 2016-09 (Actual); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Glucose tolerance assessed using a 75g-Oral Glucose Tolerance Test (OGTT) in mothers | 1 year

SECONDARY OUTCOMES:
Glycaemic and lipidic profile assessed using a fasting blood sample in children | 1 year
overweight/obesity | 1 year
  In mothers and children
abdominal obesity | 1 year
  In mothers and children
metabolic syndrome | 1 year
  In mothers and children
Breastfeeding | 1 year
  In mothers and children
Nutrition | 1 year
  In mothers and children
Physical activity | 1 year
  In mothers and children

CONTACTS AND LOCATIONS:
Overall Officials: Julie Robitaille, R.D., Ph.D., Principal Investigator — Laval University
Locations (1):
- Laval University, Institute of Nutraceuticals and Functional Foods, Québec, Canada

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Kearney M, Perron J, Marc I, Weisnagel SJ, Tchernof A, Robitaille J. Association of prenatal exposure to gestational diabetes with offspring body composition and regional body fat distribution. Clin Obes. 2018 Apr;8(2):81-87. doi: 10.1111/cob.12237. Epub 2017 Dec 13. PMID 29239129